CLINICAL TRIAL: NCT04182295
Title: Effect of Information on Placebo in the Informed Consent on the Trial Outcomes and Participant Blinding
Brief Title: Does Placebo Information Affect the Trial Outcomes and Participant Blinding?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Principal Investigator, Hyangsook Lee, KMD, PhD, Professor, Kyunghee University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KHSIRB-19-173
Record Dates: First submitted 2019-11-25; First posted 2019-12-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Muscle Soreness
Keywords: Placebo; Informed consent; Participant information leaflet; Outcome; Blinding; Sham; Acupuncture; Delayed Onset Muscle Soreness
MeSH Terms: conditions — Myalgia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- real acupuncture-full disclosure (Experimental): Participants in this group will be given real acupuncture once a day for three consecutive days including the very first visit and fully disclosed sham acupuncture information in the informed consent (i.e., fake acupuncture).
  Interventions: Device: acupuncture
- real acupuncture-partial disclosure (Experimental): Participants in this group will be given real acupuncture once a day for three consecutive days including the very first visit and partially disclosed sham acupuncture information in the informed consent (i.e., different kind of acupuncture).
  Interventions: Device: acupuncture
- sham acupuncture-full disclosure (Sham Comparator): Participants in this group will be given sham acupuncture once a day for three consecutive days including the very first visit and fully disclosed sham acupuncture information in the informed consent (i.e., fake acupuncture).
  Interventions: Device: Park Sham Needle
- sham acupuncture-partial disclosure (Sham Comparator): Participants in this group will be given sham acupuncture once a day for three consecutive days including the very first visit and partially disclosed sham acupuncture information in the informed consent (i.e., different kind of acupuncture).
  Interventions: Device: Park Sham Needle

INTERVENTIONS:
Device: acupuncture — A sterilised stainless steel needle (diameter 0.25mm X length 40mm, Dongbang Acupuncture Inc., Boryeong, Chungchenongnam-do, Korea) will be given at PC3, LI4, LI11, and LU5 of non-dominant arm for 15 minutes once a day for 3 days (immediately after inducing delayed onset muscle soreness (DOMS), and 2 consecutive days after inducing DOMS).
  Arms: real acupuncture-full disclosure; real acupuncture-partial disclosure
Device: Park Sham Needle — A Park Sham Needle (Meridius Medical Ltd. & DongBang Acuprime Ltd., Exeter, UK), non-penetrating sham acupuncture, will be given at two points on the belly of biceps brachii, 1 cun proximedially from LI11, and 1 cun laterally from PC3 of non-dominant arm for 15 minutes once a day for 3 days (immediately after inducing delayed onset muscle soreness (DOMS), and 2 consecutive days after inducing DOMS).
  Other Names: sham acupuncture
  Arms: sham acupuncture-full disclosure; sham acupuncture-partial disclosure

SUMMARY:
This is a randomised sham-controlled trial involving healthy volunteers to determine the effect of information on placebo, i.e., sham acupuncture, given in the informed consent, on the trial outcomes and blinding status of participants in a trial.

DETAILED DESCRIPTION:
A total of 89 healthy volunteers will be recruited and randomly allocated to one of the 4 groups at an identical ratio. Four groups differ in acupuncture and placebo information. It is summarized as follows:

1. to receive real acupuncture and to read fully disclosed sham acupuncture information (e.g., fake acupuncture) written in the informed consent
2. to receive real acupuncture and to read partially disclosed sham acupuncture information (e.g., different kind of acupuncture) written in the informed consent
3. to receive sham acupuncture (Park Sham Needle) and to read fully disclosed sham acupuncture information written in the informed consent
4. to receive sham acupuncture to read partially disclosed sham acupuncture information (e.g., different kind of acupuncture) written in the informed consent.

They will read informed consent with differently described placebo information following their allocation. After participants repeatedly lift a dumbbell with their non-dominant arm to induce delayed onset muscle soreness (DOMS) in their biceps brachii, they are given allocated acupuncture treatment once a day for three consecutive days including the very first visit to compare outcomes (i.e., relief of DOMS measured with pressure pain threshold and visual analogue scale) and blinding property (the participants will be asked 'which type of acupuncture do you think you have received?' and choose 1 answer out of real, sham, or don't know options).

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* not participating in other studies at the time of study participation
* voluntary participation

Exclusion Criteria:

* resistance training for more than 6 months
* experience of fracture of any of four limbs
* pregnancy or breast-feeding at the time of study participation
* analgesics within 24 hours before participation
* any other diseases or conditions that might prevent the participant from receiving acupuncture

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
the change in muscle discomfort from baseline, i.e., immediately after being induced DOMS, measured by visual analogue scale (VAS) | day 0; day 1; day 2
  Muscle discomfort of DOMS induced arm is evaluated with VAS ranging from 0 to 10 cm (with 0 indicating no discomfort and 10 experiencing the worst imaginable muscle discomfort.)
Blinding property | day 2
  Blinding property is evaluated: participants will be asked 'which type of acupuncture do you think you have received?' and choose 1 answer out of experimental group, control group, and do not know. It is calculated following the way of Bang's Blind Index; -1 indicates opposite guessing; 0 indicates random guessing; 1 indicates correct guessing.
the change in Pressure Pain Threshold (PPT) from baseline, i.e., before being induced DOMS | day 0; day 1; day 2
  Pressure Pain Threshold (PPT) will be evaluated on the 5 points of upper non-dominant arm. Five points are selected from 6 equidistance from origin to insertion of biceps brachii with an exception of the first and last point, perpendicular to the belly of the biceps brachii. Pressure was applied to each of these points with increasing force at a rate of approximately 10 N/cm2*sec until the participant reported a painful sensation, and the force value was recorded (N/cm2). An upper limit of PPt was set 50 N/cm2 to avoid bruising.

SECONDARY OUTCOMES:
Acupuncture sensation measured by De-qi questionnaire | day 0; day 1; day 2
  De-qi questionnaire (Kim et al.) is used to evaluate acupuncture sensation measured in VAS ranging from 0 to 10 cm (with 0 indicating no feeling of respective 18 items included in the questionnaire and 10 experiencing the worst imaginable feeling of respective 18 items included in the questionnaire.)

OTHER OUTCOMES:
Acupuncture credibility | day 0; day 2
  Credibility of the acupuncture treatment is evaluated using a credibility test by Vincent et al. It is a 4-item self report on a 6-point Likert scale; its score ranges from 4 to 24 point; higher score indicates more credibility over acupuncture.
Acupuncture Belief Scale (ABS) | day 0
  A Korean version of Acupuncture Belief Scale (ABS), a 36-item self-report on a 5-point Likert scale will be used to evaluate acupuncture experiences and beliefs. Its score ranges from 36 to 180 and higher score is considered more positive attitude toward acupuncture.
State-Trait Anxiety Inventory-X (STAI-X) | day 0
  A Korean version of State-Trait Anxiety Inventory-X (STAI-X); each item of anxiety has its own 20 different questions on a 4-point Likert scale. The score ranges from 20 to 80, with higher score correlating with greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Hyangsook Lee, Doctor, Principal Investigator — Kyunghee University
Locations (1):
- Acupuncture & Meridian Science Research Centre, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bang H, Ni L, Davis CE. Assessment of blinding in clinical trials. Control Clin Trials. 2004 Apr;25(2):143-56. doi: 10.1016/j.cct.2003.10.016. PMID 15020033
- [Background] Bishop FL, Adams AE, Kaptchuk TJ, Lewith GT. Informed consent and placebo effects: a content analysis of information leaflets to identify what clinical trial participants are told about placebos. PLoS One. 2012;7(6):e39661. doi: 10.1371/journal.pone.0039661. Epub 2012 Jun 27. PMID 22761859
- [Background] Cheon S, Park HJ, Chae Y, Lee H. Does different information disclosure on placebo control affect blinding and trial outcomes? A case study of participant information leaflets of randomized placebo-controlled trials of acupuncture. BMC Med Res Methodol. 2018 Jan 18;18(1):13. doi: 10.1186/s12874-018-0474-1. PMID 29347917
- [Background] Gillon R. Ethics needs principles--four can encompass the rest--and respect for autonomy should be "first among equals". J Med Ethics. 2003 Oct;29(5):307-12. doi: 10.1136/jme.29.5.307. PMID 14519842
- [Background] Harris J. In praise of unprincipled ethics. J Med Ethics. 2003 Oct;29(5):303-6. doi: 10.1136/jme.29.5.303. PMID 14519841
- [Result] Corder KE, Newsham KR, McDaniel JL, Ezekiel UR, Weiss EP. Effects of Short-Term Docosahexaenoic Acid Supplementation on Markers of Inflammation after Eccentric Strength Exercise in Women. J Sports Sci Med. 2016 Feb 23;15(1):176-83. eCollection 2016 Mar. PMID 26957941
- [Result] Dennehy EB, Webb A, Suppes T. Assessment of beliefs in the effectiveness of acupuncture for treatment of psychiatric symptoms. J Altern Complement Med. 2002 Aug;8(4):421-5. doi: 10.1089/107555302760253612. PMID 12230902
- [Result] Fleckenstein J, Niederer D, Auerbach K, Bernhorster M, Hubscher M, Vogt L, Banzer W. No Effect of Acupuncture in the Relief of Delayed-Onset Muscle Soreness: Results of a Randomized Controlled Trial. Clin J Sport Med. 2016 Nov;26(6):471-477. doi: 10.1097/JSM.0000000000000259. PMID 26540600
- [Result] Fleckenstein J, Simon P, Konig M, Vogt L, Banzer W. The pain threshold of high-threshold mechanosensitive receptors subsequent to maximal eccentric exercise is a potential marker in the prediction of DOMS associated impairment. PLoS One. 2017 Oct 6;12(10):e0185463. doi: 10.1371/journal.pone.0185463. eCollection 2017. PMID 28985238
- [Result] Graves JE, Pollock ML, Leggett SH, Braith RW, Carpenter DM, Bishop LE. Effect of reduced training frequency on muscular strength. Int J Sports Med. 1988 Oct;9(5):316-9. doi: 10.1055/s-2007-1025031. PMID 3246465
- [Result] Hubscher M, Vogt L, Bernhorster M, Rosenhagen A, Banzer W. Effects of acupuncture on symptoms and muscle function in delayed-onset muscle soreness. J Altern Complement Med. 2008 Oct;14(8):1011-6. doi: 10.1089/acm.2008.0173. PMID 18990049
- [Result] Kam-Hansen S, Jakubowski M, Kelley JM, Kirsch I, Hoaglin DC, Kaptchuk TJ, Burstein R. Altered placebo and drug labeling changes the outcome of episodic migraine attacks. Sci Transl Med. 2014 Jan 8;6(218):218ra5. doi: 10.1126/scitranslmed.3006175. PMID 24401940
- [Result] Lin MJ, Nosaka K, Ho CC, Chen HL, Tseng KW, Ratel S, Chen TC. Influence of Maturation Status on Eccentric Exercise-Induced Muscle Damage and the Repeated Bout Effect in Females. Front Physiol. 2018 Jan 5;8:1118. doi: 10.3389/fphys.2017.01118. eCollection 2017. PMID 29354073
- [Result] Myers MG, Cairns JA, Singer J. The consent form as a possible cause of side effects. Clin Pharmacol Ther. 1987 Sep;42(3):250-3. doi: 10.1038/clpt.1987.142. PMID 3621780
- [Result] Shimano T, Kraemer WJ, Spiering BA, Volek JS, Hatfield DL, Silvestre R, Vingren JL, Fragala MS, Maresh CM, Fleck SJ, Newton RU, Spreuwenberg LP, Hakkinen K. Relationship between the number of repetitions and selected percentages of one repetition maximum in free weight exercises in trained and untrained men. J Strength Cond Res. 2006 Nov;20(4):819-23. doi: 10.1519/R-18195.1. PMID 17194239
- [Result] Webster RK, Weinman J, Rubin GJ. Positively Framed Risk Information in Patient Information Leaflets Reduces Side Effect Reporting: A Double-Blind Randomized Controlled Trial. Ann Behav Med. 2018 Oct 22;52(11):920-929. doi: 10.1093/abm/kax064. PMID 30346496